CLINICAL TRIAL: NCT06495996
Title: PROTECTOR: Evaluating the Safety and Effectiveness of the Protrieve Sheath in Preventing Clinically Significant Intraprocedural Pulmonary Embolism by Providing Embolic Protection in the IVC During Thrombectomy Procedures to Treat DVT
Brief Title: The Protrieve PROTECTOR Study
Acronym: PROTECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-003
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis
Keywords: Venous Thromboembolism; Deep Venous Thrombosis; Percutaneous Mechanical Thrombectomy
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Protrieve Sheath (Experimental): The Protrieve Sheath is intended for embolic protection in the inferior vena cava (IVC) to prevent clinically significant intraprocedural pulmonary embolism during mechanical thrombectomy procedures in patients with high risk of embolization.
  Interventions: Device: Percutaneous mechanical thrombectomy (PMT)

INTERVENTIONS:
Device: Percutaneous mechanical thrombectomy (PMT) — Percutaneous mechanical thrombectomy (PMT) is the endovascular removal of thrombus by catheter-based mechanical or aspiration methods. The term PMT generally describes interventional procedures performed without the use of lytic agents and frequently involves instrumentation in extensive amounts of fresh thrombus.

SUMMARY:
The Protrieve PROTECTOR Study is a prospective, single-arm, multicenter study of the Protrieve Sheath.

DETAILED DESCRIPTION:
The primary study objective is to evaluate the safety and effectiveness of the Protrieve Sheath in preventing clinically significant intraprocedural pulmonary embolism by providing embolic protection in the IVC during thrombectomy procedures to treat DVT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Planned intervention for DVT presenting with one or more of the following characteristics indicative of elevated risk for PE:

   1. Bilateral iliofemoral DVT
   2. Clot extending into or located in the IVC
   3. In-stent thrombosis
   4. Presence of thrombosed IVC filter
   5. Other features that the investigator deems put the subject at elevated risk for thromboembolism
3. Willing and able to provide informed consent

Exclusion Criteria:

1. Current symptomatic PE
2. Known anatomic inability to place Protrieve device via jugular vein access site
3. Presence of clot extending to the IVC-Right Atrial junction or in the SVC
4. Subject is pregnant
5. Severe allergy to iodinated contrast agents that cannot be mitigated
6. INR > 1.7 if not currently on anticoagulation therapy, platelets < 50,000/μl which cannot be corrected prior to enrollment, or Hemoglobin < 8.0 g/dL
7. Severe renal impairment in patients who are not yet on dialysis that in the Investigator's discretion would pose risk to the patient with the use of marketed contrast agents
8. Subject is participating in another study that may interfere with this study
9. Subject has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject
10. Subject has previously completed or withdrawn from this study
11. Limb-threatening circulatory compromise (e.g., phlegmasia)
12. Uncontrolled severe hypertension on repeated readings (systolic > 180mmHg or diastolic > 105mmHg)
13. Severe allergy, hypersensitivity to, or thrombocytopenia from heparin
14. Inability to provide therapeutic anticoagulation per Investigator discretion
15. Known hypercoagulable states that, in the opinion of the Investigator, cannot be medically managed throughout the study period
16. Inability to be a candidate for intervention due to medical or technical reasons based on physician judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Measure: | 24 Hours (+-12 Hours)
  a. Clinically significant PE
Primary Safety Measure: | 24 Hours (+-12 Hours)
  1. Protrieve device-related Major Adverse Events (MAEs)
  2. Major Protrieve access site complications

SECONDARY OUTCOMES:
Capture of Thromboembolic Material | 24 Hours (+-12 Hours)
  a. Capture and removal of thromboembolic material in the Protrieve funnel, as assessed by proportion of study cases where any material was either entrapped in the funnel or removed via Protrieve
Device Success | 24 Hours (+-12 Hours)
  b. Device success, defined as successful delivery, deployment, and retrieval of the Protrieve device without complications
Venous Access Routes | 24 Hours (+-12 Hours)
  c. Thrombectomy via supplementary venous access routes
Estimated Percentage of the Protrieve Funnel Obstructed | 24 Hours (+-12 Hours)
  d. Estimated percentage of the Protrieve funnel obstructed by clot, as observed by visual inspection or imaging
Blood Transfusions | 24 Hours (+-12 Hours)
  e. Blood transfusions associated with Protrieve Sheath access site bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Sabah D Butty, MD, Principal Investigator — Indiana University Health Methodist Hospital
Locations (15):
- United States (15):
  - Hoag Hospital, Newport Beach, California
  - Yale University, New Haven, Connecticut
  - Baptist Health South Florida, Miami, Florida
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University Medical Center Southern Nevada, Las Vegas, Nevada
  - Englewood Hospital, Englewood, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No